CLINICAL TRIAL: NCT04685005
Title: Double Blind Placebo and Active (Caffeine) Controlled Study to Examine the Effects of 3 Doses of "WakeUp" Herbal Beverage Containing Green Tea (Instead of Ginkgo Biloba) on Vigilance and Function of Healthy Volunteers Following Lunch
Brief Title: "WakeUp" for Vigilance Following Lunch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Giora Pillar, MD, PhD, Head of Department of Pediatrics and Sleep Clinic, Carmel Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WU 2018 GT
Record Dates: First submitted 2020-12-07; First posted 2020-12-28 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Wuc protein, Drosophila; Caffeine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized regarding the order of the various beverages they drink, in a double blind placebo and active control model.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be kept by the manufacturer of the beverages (Frutarom USA, Inc). All 5 beverages (placebo, 100mg Caffeine, WakeUp® regular dose, WakeUp® double dose, and WakeUp® triple dose) will be marked by a letter beween A to E, which will be blinded to the participants and the staff of the study. Only after the completion of the study (all 30 participants), and statistical analysis and reporting will the various beverages (letters) will be unblinded. The only occasion of unblinding prior to study completion will be the unexpected occasion of a serious side effect.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Wake up (Experimental): Drinking regular formula of Wake Up
  Interventions: Dietary Supplement: "Wake Up"; Dietary Supplement: Caffeine
- Caffeine (Active Comparator): Drinking 100mg of Caffeine
  Interventions: Dietary Supplement: "Wake Up"; Dietary Supplement: Caffeine
- Placebo (Placebo Comparator): Drinking Placebo (only water with sugar)
  Interventions: Dietary Supplement: "Wake Up"; Dietary Supplement: Caffeine
- Wake up Double Dose (Experimental): Drinking formula of Wake Up with double doses of guarana, green tea, elderberry and Fruit-up
  Interventions: Dietary Supplement: "Wake Up"; Dietary Supplement: Caffeine
- Wake up tripple dose (Experimental): Drinking formula of Wake Up with tripple doses of guarana, green tea, elderberry and Fruit-up
  Interventions: Dietary Supplement: "Wake Up"; Dietary Supplement: Caffeine

INTERVENTIONS:
Dietary Supplement: "Wake Up" — The current composition of the WakeUp® beverage consists of herbal extracts of guarana, green tea, elderberry and Fruit-up
  Other Names: Caffeine, Placebo
Dietary Supplement: Caffeine — Caffeine

SUMMARY:
This is a single center, double-blind, placebo and active controlled clinical trial comprised of a single drink of WakeUp beverage (in 3 doses) compared to Caffeine (100mg) and placebo given to health volunteers.

Participants will be randomized regarding the order of the various beverages. Healthy volunteers or stable (under treatment) patients with chronic diseases) will be included. They will be studied 5 times, in a 2-14 days period, each time during noontime (between 11:30 and 15:00).

Each day of the study, the participants will follow the following schedule:

Lunch any time between 11:30 and 13:30 Time 0: Immediately after lunch a baseline set of assessment. Time 30min: Participants will then consume a beverage (which will be either placebo or 100mg caffeine or single/double/triple dose of WakeUp in the various days) Time 60min: Repeat the same set of assessments as done 30min after beverage Time 150min: Repeat the same set of assessments 2 hours after beverage Time 180min: End of day assessment

DETAILED DESCRIPTION:
This is a randomized, double-blind, controlled study with placebo and active control, to test the efficacy and safety of WakeUp on alertness and function in 30 healthy or chronically ill but stable adult volunteers.

Participants and recruitment Thirty volunteers will be recruited via advertisements (in the hospital and university environment). Initial assessment of inclusion and exclusion criteria will take place on the primary visit, and once participants have met the criteria for participation and sign an informed consent, they will enter the study and undergo randomization. It is permitted for participants to have any chronic disease (such as hypertension or diabetes) if they are stable and controlled. Participants will continue taking their own medications (as long as they are not stimulants or sedating, in which case the subject will be excluded).

Study procedure and schedule This is a single center, double-blind, placebo and active controlled clinical trial comprised of a single drink of WakeUp® beverage (in 3 doses) compared to caffeine (100mg) and placebo given to health volunteers. Participants will be randomized regarding the order of the various beverages.

The following visits and schedule will comprise the study:

1. Screening visit: In this visit study procedures will be expained, inclusionqexclusion criteria determined, informed consent signed).
2. Visit 1: Participants eats their regular lunce following which a first set of studies takes place (see below). Immediately thereafter the participant drinks the tested beverage (marked A, B, C, D, E or F, randomized order regarding which beverage of the 6 is drank at each specific study day, blinded to the participant and the staff). Thirty minutes after drinking a second set of studies will take place (exactly equal to the previous set of studies). A third set of studies (exactly the same as the previous two) will take place 2 hours following the drink.
3. Visits 2, 3, 4, and 5 are exactly like visit 1, just that the beverage is one of the others (randomized), such that each participants after completing 5 visits had all tested beverages: placebo, 100mg Caffeine, WakeUp® regular dose, WakeUp® double dose, WakeUp® triple dose.
4. Visit 7: A telephone call or a face-to-face visit (based on the preference of the participants) one week after the study to make sure there are no side effects and to close participation.

The time between screening and visit 1 can be any time between 0 (screening and visit 1 on the same day) to 1 month.

The time between any two other visits (visit 1 to 2, 2 to 3 etc) can be any time between 1 to 14 days.

Each one of visits 1 to 5 will begin after lunch, between 11:30 and 15:00, preferable at the same time in all visits 1 to 5.

Randomization Treatment will be randomized for the order of beverage tested (A to E) in visits 1 to 5 by a computer-generated randomization scheme (randome function written in JAVA). At the beginning of visit 1 randomization will be performed for the whole study period (i.e. for which of beverages A,B,C,D,E to be drunk on which of the visits 1,2,3,4,5).

Blinding Blinding will be kept by the manufacturer of the beverages (Frutarom USA, Inc). All 5 beverages (placebo, 100mg Caffeine, WakeUp® regular dose, WakeUp® double dose, and WakeUp® triple dose) will be marked by a letter beween A to E, which will be blinded to the participants and the staff of the study. Only after the completion of the study (all 30 participants), and statistical analysis and reporting will the various beverages (letters) will be unblinded. The only occasion of unblinding prior to study completion will be the unexpected occasion of a serious side effect.

Set of testing for the study

At all testing times (3 times at every visit from visit 1 to 5, each time point after lunch, 30min after beverage, 2h after beverage) the following tests will be performed:

Vital signs (blood pressure and pulse rate) Asking about side effects Visual Analog Scale for Alertness (see above) Immediate word recall test (see above) Neurocognitive function testing by Cambridge Cognition on an ipad tablet.

The following neurocognitive function tests will be performed:

Attention:

RTI- Reaction Time - 2-3 minutes

The participant must select and hold a button at the bottom of the screen. Circles are presented above (one for the simple mode, and five for the five-choice mode.) In each case, a yellow dot will appear in one of the circles, and the participant must react as soon as possible, releasing the button at the bottom of the screen, and selecting the circle in which the dot appeared. Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.

RVP - Rapid Visual Information Processing - 7 minutes

A white box is shown in the centre of the screen, inside which digits from 2 to 9 appear in a pseudo-random order, at the rate of 100 digits per minute. Participants are requested to detect target sequences of digits (for example, 2-4-6, 3-5-7, 4-6-8). When the participant sees the target sequence they must respond by selecting the button in the centre of the screen as quickly as possible. The level of difficulty varies with either one- or three-target sequences that the participant must watch for at the same time. Outcome measures cover latency (speed of response), probability of false alarms and sensitivity.

Executive Function:

MTT- Multitasking Test- 8 minutes

The test displays an arrow which can appear on either side of the screen (right or left) and can point in either direction (to the right or to the left). Each trial displays a cue at the top of the screen that indicates to the participant whether they have to select the right or left button according to the "side on which the arrow appeared" or the "direction in which the arrow was pointing". In some sections of the task this rule is consistent across trials (single task) while in others it may change from trial to trial in a randomised order (multitasking). Using both rules in a flexible manner places a higher demand on cognition than using a single rule.

Some trials display congruent stimuli (e.g. arrow on the right side pointing to the right) whereas other trials display incongruent stimuli, which require a higher cognitive demand (e.g. arrow on the right side of the screen pointing to the left). Outcome measures for the Multitasking Test include response latencies and error scores that reflect the participant's ability to manage multitasking and the interference of incongruent task-irrelevant information on task performance (i.e. a Stroop-like effect).

SSP- Spacial Span - 5 minutes

White squares are shown on the screen, some of which briefly change colour in a variable sequence. The participant must then select the boxes which changed colour in the same order that they were displayed by the computer (for the forward variant) or in the reverse order (for backward variant). The number of boxes in the sequence increases from two at the start of the test, to nine at the end and the sequence and colour are varied through the test. Outcome measures cover span length (the longest sequence successfully recalled), errors, number of attempts and latency (speed of response).

Memory:

SWM-Spatial Working Memory - 4 minutes

The test begins with a number of coloured squares (boxes) shown on the screen. The aim of this test is that by selecting the boxes and using a process of elimination, the participant should find one yellow 'token' in each of a number of boxes and use them to fill up an empty column on the right-hand side of the screen. Depending on the difficulty level used for this test, the number of boxes can be gradually increased until a maximum of 12 boxes are shown for the participants to search. The colour and position of the boxes used are changed from trial to trial to discourage the use of stereotyped search strategies. Outcome measures include errors (selecting boxes that have already been found to be empty and revisiting boxes which have already been found to contain a token) and strategy and latency.

The data for vital signs, potential side effects, alertness and iWRT will be kept in a local case report form. The data of the Cambridge Cognition tests are stored in the tablet, or sent to the cloud if the tablet is connected to wifi at that time. All data are sent to the cloud whenever the tablet connects to wifi. The data are compiled by Cambridge and the raw data are put into a CSV file which can be downloaded from the tablet directly and can open in Microsoft Excel. The secure private cloud environment is provided by HIPAA-accredited supplier Armor. The data are secured via military grade encryption (256-bit key file encryption) and are only accessible to authorized users. As an additional security measure, Cambridge Cognition commissions an independent security check on the system each year and Cambridge Cognition and the CANTAB Connect platform have been audited by the Medicines and Healthcare products Regulatory Agency and British Standards Institute, as well as external audits arranged by customers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers or chronically ill patients in stable condition
2. Adults age 18 and above
3. Volunteers who are willing and able to sign the informed consent

Exclusion Criteria:

1. Children aged less than 18 years.
2. Subjects participating in another study
3. Subjects who are unable to comply with the study procedures.
4. Patients in an unstable medical condition.
5. Patients who are treated with sedating or stimulant medications
6. Subjects who have taken a dietary supplement within one week of the study initiation
7. Subjects who have drunk or eaten any caffeine-containing beverage or food after 7:00 in the morning of any test day
8. Any reason that, in the opinion of the investigator, may make the subject unfit for this clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Alertness assessed at baseline before drinking Wake Up | time 0 - baseline
  measured by neurocognitive functional test assessed by reaction time response for five-choice variants - a test by Cambridge Cognition company, performed on an iPad tablet
Alertness assessed at 30 minutes after drinking Wake Up | 30 minutes
  measured by neurocognitive functional test assessed by reaction time response for five-choice variants - a test by Cambridge Cognition company, performed on an iPad tablet
Alertness assessed at 120 minutes after drinking Wake Up | 120 minutes
  measured by neurocognitive functional test assessed by reaction time response for five-choice variants - a test by Cambridge Cognition company, performed on an iPad tablet

SECONDARY OUTCOMES:
Neurocognitive attention test at baseline before drinking Wake Up | time 0 - baseline
  by Tablet Tests: attention test provided by Cambridge Cognition
Neurocognitive attention test at 30 minutes after drinking Wake Up | 30 minutes
  by Tablet Tests: attention test provided by Cambridge Cognition
Neurocognitive attention test at 120 minutes after drinking Wake Up | 120 minutes
  by Tablet Tests: attention test provided by Cambridge Cognition
Neurocognitive executive function test at baseline before drinking Wake Up | time 0 - baseline
  by Tablet Tests: executive function test provided by Cambridge Cognition
Neurocognitive executive function test at 30 minutes after drinking Wake Up | 30 minutes
  by Tablet Tests: executive function test provided by Cambridge Cognition
Neurocognitive executive function test at 120 minutes after drinking Wake Up | 120 minutes
  by Tablet Tests: executive function test provided by Cambridge Cognition
Neurocognitive memory test at baseline before drinking Wake Up | time 0 - baseline
  by Tablet Tests: memory test provided by Cambridge Cognition
Neurocognitive memory test at 30 minutes after drinking Wake Up | 30 minutes
  by Tablet Tests: memory test provided by Cambridge Cognition
Neurocognitive memory test at 120 minutes after drinking Wake Up | 120 minutes
  by Tablet Tests: memory test provided by Cambridge Cognition

CONTACTS AND LOCATIONS:
Overall Officials: Giora P Pillar, Prof, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
The data are stored in the tablet, or sent to the cloud if the tablet is connected to wifi at that time. All data are sent to the cloud whenever the tablet connects to wifi. The data are compiled by Cambridge and the raw data are put into a CSV file which can be downloaded from the tablet directly and can open in Microsoft Excel. The secure private cloud environment is provided by HIPAA-accredited supplier Armor. The data are secured via military grade encryption (256-bit key file encryption) and are only accessible to authorized users. As an additional security measure, Cambridge Cognition commissions an independent security check on the system each year. In addition, Cambridge Cognition and the CANTAB Connect platform have been audited by the Medicines and Healthcare products Regulatory Agency and British Standards Institute, as well as via external audits arranged by customers.